CLINICAL TRIAL: NCT07259941
Title: PET-CT Imaging Findings and Metabolic Parameters in Elderly Patients With Lymphoma
Brief Title: PET-CT in Lymphoma Among the Eldery
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mamdouh Ekram, Resident at Nuclear Medicine unit, Radiotherapy and Nuclear Medicine Department, South Egypt Cancer Institute, Assiut University
Other Study IDs: PET-CT Imaging in Lymphoma
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: PET-CT; Lymphoma; Elderly; Metabolic Parameters
Keywords: PET-CT; Lymphoma; Elderly; metabolic parameters
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
This study investigates PET-CT imaging patterns and metabolic parameters in elderly patients (≥60 years) diagnosed with lymphoma, aiming to enhance diagnostic accuracy and prognosis using 18F-FDG PET/CT scans.

DETAILED DESCRIPTION:
This cross-sectional study involves both retrospective and prospective data collection from elderly lymphoma patients (aged 60 years or older) at the Nuclear Medicine Unit, South Egypt Cancer Institute. It evaluates the PET-CT imaging findings alongside metabolic parameters such as Standardized Uptake Value (SUV), Metabolic Tumor Volume (MTV), and Total Lesion Glycolysis (TLG). The study addresses diagnostic challenges in elderly patients due to atypical presentations and comorbidities and fills the gap of scarce local data in Egypt. Imaging analysis includes visual and semiquantitative assessment of lymphatic and extranodal lesions post-injection of 18F-FDG, assessing tumor metabolic activity to provide prognostic insights. Data analysis uses SPSS with relevant statistical tests to validate findings.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 60 years

Histopathological diagnosis of lymphoma

Exclusion Criteria:

- Presence of other concurrent active malignancies

Uncontrolled diabetes mellitus with blood glucose > 200 mg/dL at the time of PET/CT scan

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants include elderly patients (≥60 years) with confirmed lymphoma diagnosis through histopathological examination. Excluded are individuals with other active cancers or uncontrolled diabetes mellitus (blood glucose > 200 mg/dL), which could interfere with PET scan accuracy. Patients must have fasting blood glucose < 200 mg/dL before 18F-FDG injection and are prepared per standardized protocols. The sample size is calculated to be approximately 63 patients, providing adequate statistical power based on confidence limits and previous positive PET findings in elderly lymphoma cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
FDG-PET/CT Imaging Pattern Description in Elderly Lymphoma Patients | At time of initial PET/CT scan performed as part of routine clinical evaluation
  The main outcome is the characterization of metabolic and anatomical findings from 18F-FDG PET/CT scans among elderly patients (≥60 years) diagnosed with lymphoma. This includes describing the visual appearance, extent, and distribution of disease lesions observed on initial imaging.